CLINICAL TRIAL: NCT03102554
Title: Utilizing Whole Exome Sequencing and Genomics to Improve Our Understanding of Differences of Sex Development (DSD) and Hypospadias
Brief Title: Genetics of Differences of Sex Development and Hypospadias
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Yee-Ming Chan, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00012912
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Disorders of Sex Development; Hypospadias
Keywords: Exome Sequencing
MeSH Terms: conditions — Disorders of Sex Development; Hypospadias

STUDY DESIGN:
Intervention Model Description: Longitudinal cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genetic Testing (Experimental): Subjects will provide a DNA sample, which will be screened for variants in genes related to DSD/hypospadias. Probands/parents who wish to receive results of genetic testing related to DSD/hypospadias will receive these results directly from the research study. Parents who receive results of genetic testing for probands 17 years old or younger will complete questionnaires at the time of enrollment, right after receiving genetic results, and 3 months after receiving genetic results.
  Interventions: Genetic: Return of Genetic Results

INTERVENTIONS:
Genetic: Return of Genetic Results — The results of testing for genetic causes of DSD/hypospadias will be returned to parents of subjects who elect to receive these results.

SUMMARY:
This study seeks to identify genetic causes of conditions that affect the gonads and genitals, and to study the impact on families of receiving genetic results.

DETAILED DESCRIPTION:
This study seeks to understand the genetic causes of conditions that affect the development of the genitals, such as differences of sex development (DSD) and hypospadias, and the impact on families of receiving genetic results. The investigators are recruiting individuals with DSD and/or hypospadias without a clear genetic cause along with their family members for our research study. The investigators will collect samples for genetic studies. The investigators will review the clinical record for history, labs and physical exam information. The investigators will return results of genetic testing to parents/guardians of children with DSD/hypospadias and have them complete questionnaires to assess the impact of receiving these results.

ELIGIBILITY:
Inclusion Criteria:

* Genital or gonadal abnormalities as evidenced by physical examination or imaging (including but not limited to hypospadias, microphallus, clitoromegaly, ambiguous genitalia), with no cause identified by standard clinical evaluation

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Decision Regret | 3 months after return of genetic results
  Score on Decision Regret Scale

SECONDARY OUTCOMES:
Parenting-Related Stress | 3 months after return of genetic results compared to baseline
  Score on Parenting Stress Index
Child Health-Related Stress | 3 months after return of genetic results compared to baseline
  Score on Child Health Worry Scale
Anxiety | 3 months after return of genetic results compared to baseline
  Score on Generalized Anxiety Disorder-7
Depression | 3 months after return of genetic results compared to baseline
  Score on Patient Health Questionnaire-9
Partner Relationship | 3 months after return of genetic results compared to baseline
  Score on Kansas Marital Satisfaction Scale
Partner Blame | 3 months after return of genetic results compared to baseline
  Score on this novel measure
Stigma | baseline, 3 months after return of genetic results
  Score on Questionnaire, "Stigma Related to Having a Child with a Urogenital Condition"
Quality of Life score | baseline, 3 months after return of genetic results
  Score on Questionnaire, "Quality of Life Related to Having a Child with a Urogenital Condition"

CONTACTS AND LOCATIONS:
Overall Officials: Yee-Ming Chan, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No